CLINICAL TRIAL: NCT01444846
Title: Phase 2 Study of the Safety and Efficacy of an Oral Formulation of SPI-1005 for Prevention of Temporary Auditory Threshold Shift
Brief Title: Otoprotection With SPI-1005 for Prevention of Temporary Auditory Threshold Shift
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sound Pharmaceuticals, Incorporated (Industry)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SPI-1005-202
Record Dates: First submitted 2011-09-29; First posted 2011-10-03 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Temporary Auditory Threshold Shift
Keywords: Temporary Auditory Threshold Shift; Hearing Loss; Deafness; SPI-1005; Ebselen
MeSH Terms: conditions — Hearing Loss; Deafness | interventions — ebselen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SPI-1005 Low dose (Active Comparator): 200mg SPI-1005, capsule, bid, po, x4d
  Interventions: Drug: SPI-1005 Low dose
- SPI-1005 Middle Dose (Active Comparator): 400mg SPI-1005, capsule, bid, po, x4d
  Interventions: Drug: SPI-1005 Middle dose
- SPI-1005 High Dose (Active Comparator): 600mg SPI-1005, capsule, bid, po, x4d
  Interventions: Drug: SPI-1005 High dose
- Placebo (Placebo Comparator): 0mg SPI-1005, capsule, bid, po, x4d
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPI-1005 Low dose — Oral capsules, 200 mg ebselen, twice daily, 4 days
  Other Names: 200 mg Ebselen
  Arms: SPI-1005 Low dose
Drug: SPI-1005 Middle dose — Oral capsules, 400 mg ebselen, twice daily, 4 days
  Other Names: 400 mg Ebselen
  Arms: SPI-1005 Middle Dose
Drug: SPI-1005 High dose — Oral capsules, 600 mg ebselen, twice daily, 4 days
  Other Names: 600mgEbselen
  Arms: SPI-1005 High Dose
Drug: Placebo — Oral capsules, 0 mg ebselen, twice daily, 4 days
  Other Names: 0 mg Ebselen
  Arms: Placebo

SUMMARY:
Exposure to loud sounds can cause hearing loss. The purpose of this research study is to evaluate potential prevention of temporary changes in hearing that may occur after listening to music through an iPod or personal music player. We will measure temporary changes in hearing in subjects who listen to music and take either the study drug, SPI-1005, or a placebo for 4 days. SPI-1005 is a proprietary preparation of ebselen that allows it to be taken by mouth. Ebselen contains the mineral selenium and behaves like Glutathione Peroxidase, an enzyme that helps to rid the body of damaging chemicals caused by loud sounds.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects at the time of enrollment.
* Each subject will give informed consent to participate in this study and agrees to the treatment protocol.
* Each subject will be interviewed regarding hearing and health to reveal any history of hearing loss, tinnitus, known ear pathology, use of any potentially ototoxic medications (i.e. diuretics, minocycline).
* Non-occupational sound exposure (e.g., concerts, firearms, fireworks, power tools) will be avoided during the 24-hour period preceding baseline testing and throughout the duration of the study.
* Subjects will have vital signs (i.e., heart rate, blood pressure, respirations, temperature) within normal limits upon medical examination.
* Subjects must have normal audiologic assessment at baseline consisting of:
* Baseline audiometric evaluation confirms that subjects have symmetric hearing with air conduction thresholds no worse than 25 decibels of Hearing Loss (dBHL) at frequencies between 0.25 to 8 kilo Hertz (kHz) bilaterally.
* No significant threshold asymmetry (i.e. greater than 15 dB) between the ears at any tested frequency.
* No significant air-bone gaps (i.e. greater than 10 dB)
* Type A tympanograms bilaterally, defined as a range of -140 to +40 dekaPascals (daPa) based on the 90% range for adults (Margolis and Hunter 2000)

Exclusion Criteria:

* • Subjects with abnormal hearing levels > 25 dBHL at any tested frequency (250, 500, 1000, 2000, 3000, 4000, 6000 and 8000 Hz) for either ear.
* Exposure to any duration of non-occupational high-level sound (e.g., concerts, firearms, fireworks, power tools) during the 24 hour period preceding baseline audiometric testing as revealed in the subject questionnaire or during the medical examination.
* Pathology of the external ear discovered upon otoscopic examination.
* Pathology of the middle ear revealed by otoscopic examination, abnormal tympanometry, or reported history of middle ear problems.
* Pathology of the inner ear or auditory nerve as revealed by reported history.
* Subject complaints of aural pain, pressure, fullness, or drainage.
* Subjects testing positive for pregnancy will be excluded from the study.
* Subjects with other medical/health issues that would preclude voluntary participation in a drug study may be excluded at the discretion of the Principal Investigator.
* Subjects that have previously received any known potentially ototoxic medication. This includes, but is not limited to, high dose salicylates (>2 g/day), platinum-based chemotherapeutics and aminoglycoside antibiotics, such as streptomycin, gentamicin,tobramycin, amikacin, neomycin, and netilmycin.
* Subjects that are currently using of any potentially ototoxic medications (i.e. diuretics or minocycline).
* Subjects that have received any investigational treatment (drug or device) in the six months prior to this study.
* Subjects exhibiting or self-reporting shortness of breath, wheezing, coughing, or hemoptysis

Ages: 18 Years to 31 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Reduction in Temporary Threshold Shift | 1 week
  Post-sound exposure pure tone audiometry will be compared with baseline (i.e., immediately pre-sound exposure) testing to determine group mean level hearing threshold shift changes between treated and placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Le Prell, PhD, Principal Investigator — University of Florida; Jonathan Kil, MD, Study Director — Sound Pharmaceuticals, Inc; Eric D Lynch, PhD, Study Director — Sound Pharmaceuticals, Inc
Locations (1):
- University of Florida, Gainsville, Florida, United States

REFERENCES:
- [Background] Pourbakht A, Yamasoba T. Ebselen attenuates cochlear damage caused by acoustic trauma. Hear Res. 2003 Jul;181(1-2):100-8. doi: 10.1016/s0378-5955(03)00178-3. PMID 12855368
- [Background] Lynch ED, Gu R, Pierce C, Kil J. Ebselen-mediated protection from single and repeated noise exposure in rat. Laryngoscope. 2004 Feb;114(2):333-7. doi: 10.1097/00005537-200402000-00029. PMID 14755214
- [Background] Lynch ED, Gu R, Pierce C, Kil J. Reduction of acute cisplatin ototoxicity and nephrotoxicity in rats by oral administration of allopurinol and ebselen. Hear Res. 2005 Mar;201(1-2):81-9. doi: 10.1016/j.heares.2004.08.002. PMID 15721563
- [Background] Yamasoba T, Pourbakht A, Sakamoto T, Suzuki M. Ebselen prevents noise-induced excitotoxicity and temporary threshold shift. Neurosci Lett. 2005 Jun 3;380(3):234-8. doi: 10.1016/j.neulet.2005.01.047. Epub 2005 Feb 1. PMID 15862892
- [Background] Lynch ED, Kil J. Compounds for the prevention and treatment of noise-induced hearing loss. Drug Discov Today. 2005 Oct 1;10(19):1291-8. doi: 10.1016/S1359-6446(05)03561-0. PMID 16214673
- [Background] Kil J, Pierce C, Tran H, Gu R, Lynch ED. Ebselen treatment reduces noise induced hearing loss via the mimicry and induction of glutathione peroxidase. Hear Res. 2007 Apr;226(1-2):44-51. doi: 10.1016/j.heares.2006.08.006. Epub 2006 Oct 6. PMID 17030476
- [Background] Lynch E, Kil J. Development of Ebselen, a Glutathione Peroxidase Mimic, for the Prevention and Treatment of Noise-Induced Hearing Loss. Semin Hear 2009; 30(1): 047-055
- [Background] Le Prell CG, Yang Q, Harris JG. Modification of digital music files for use in human temporary threshold shift studies. J Acoust Soc Am. 2011 Oct;130(4):EL142-6. doi: 10.1121/1.3630017. PMID 21974483
- [Background] Le Prell CG, Dell S, Hensley B, Hall JW 3rd, Campbell KC, Antonelli PJ, Green GE, Miller JM, Guire K. Digital music exposure reliably induces temporary threshold shift in normal-hearing human subjects. Ear Hear. 2012 Nov-Dec;33(6):e44-58. doi: 10.1097/AUD.0b013e31825f9d89. PMID 22885407
- [Derived] Kil J, Lobarinas E, Spankovich C, Griffiths SK, Antonelli PJ, Lynch ED, Le Prell CG. Safety and efficacy of ebselen for the prevention of noise-induced hearing loss: a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet. 2017 Sep 2;390(10098):969-979. doi: 10.1016/S0140-6736(17)31791-9. Epub 2017 Jul 14. PMID 28716314
- [Derived] Spankovich C, Le Prell CG. Associations between dietary quality, noise, and hearing: data from the National Health and Nutrition Examination Survey, 1999-2002. Int J Audiol. 2014 Nov;53(11):796-809. doi: 10.3109/14992027.2014.921340. Epub 2014 Jun 30. PMID 24975234